CLINICAL TRIAL: NCT05615740
Title: Prevention of Onset and Transition to an Advanced Form of Diabetic Retinopathy in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 03_RVO-FNOs_2022
Record Dates: First submitted 2022-10-27; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; optical coherence tomography; fluorescein angiography; diabetes mellitus
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled into two groups - healthy pediatric population and children with diabetes mellitus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy pediatric patients (Active Comparator): Healthy pediatric patients will undergo optical coherence tomography.
  Interventions: Diagnostic Test: Optical coherence tomography (OCTA)
- Children with diabetes mellitus (Active Comparator): Children with diabetes mellitus will undergo optical coherence tomography.
  Interventions: Diagnostic Test: Optical coherence tomography (OCTA)

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography (OCTA) — OCTA can detect the passage of individual blood elements (mostly erythrocytes) through capillaries and larger vessels in real-time

SUMMARY:
The primary goal of the project is to create a normative database from data collected from a healthy pediatric population. A secondary aim is to compare normative data with data from pediatric patients with pre-existing type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Diabetic retinopathy, or damage to the retina caused by diabetes, is one of the most common complications in all patients with newly diagnosed diabetes mellitus of both types. These are mainly pathological changes affecting the vascular supply of the retina, which precede changes affecting the peripheral nervous system.

Children and in general patients with type I diabetes mellitus are around 0.6% of the population in the long term. the first changes in the retinal vessels can usually be expected after 2-5 years from the first detection of the disease. These changes are diagnosed using a biomicroscopic examination of the fundus.

Until recently, the only possible examination method was fluorescein angiography (FAG). It is an invasive examination with a fluorescein solution administered into a peripheral vein through a cannula and further photo documentation of the flow dynamics through the vascular bed in blue (cobalt) light. The flow time in individual phases of filling is recorded.

The disadvantage is the necessary cooperation of the child, the need to establish peripheral venous access, the risk of an allergic reaction to the contrast material, and the duration of the examination lasting two or more hours.

These disadvantages disappeared with the advent of optical coherence tomography and the angiographic mode - OCTA.

OCTA can detect the passage of individual blood elements (mostly erythrocytes) through capillaries and larger vessels in real-time and thus compile maps of individual vascular networks in the retina and choroid. The advantage is that the examination is not invasive, it is not necessary to inject a dye into the patient's bloodstream and no special preparation is required. The device is classified as a Class 1 laser, which is safe for the human eye. The examination is not painful or uncomfortable.

Due to the relatively short period of use in practice, there is still a lack of data from findings in a healthy population. In the past, normative databases of adult patients were compiled for comparing the state of the healthy central area of the eye using OCTA. Data for the child population, especially the Central European one, is missing or has been collected on a small sample only.

The primary goal of the project is to create a normative database from data collected from a healthy pediatric population. A secondary aim is to compare normative data with data from pediatric patients with pre-existing type 1 diabetes mellitus.

It is anticipated that 100-150 children aged 6-15 will be enrolled at the Centre for Visually Impaired Children of the University of Ostrava as part of regular check-ups. Depending on the degree of cooperation of the child, the examination takes around two minutes.

ELIGIBILITY:
Inclusion Criteria:

* emmetropia
* slight refractive error
* best-corrected visual acuity equal to or better than 6/6 Schnellen optotypes

Exclusion Criteria:

* general disease that by its nature affects or can affect the retina and the vascular system of the eye
* concomitant vascular or other retinal diseases

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Vascular density in central and peripheral retina - healthy subjects | 3 years
  The primary goal of the project is measurement of vascular density in central and peripheral retina in healthy subjects using OCT Spectralis (Heidelberg Engineering, Germany). Vascular density is ratio between areas with and without vascular tissue. Data will be analysed by ImageJ software (National Institutes of Health, USA). Normative data will be collected from healthy individuals 6-15 years old.

SECONDARY OUTCOMES:
Vascular density in central and peripheral retina - diabetic patients | 3 years
  The secondary goal of the project is measurement of vascular density in central and peripheral retina in diabetic patients using OCT Spectralis (Heidelberg Engineering, Germany). Data will be analysed by ImageJ software (National Institutes of Health, USA). Normative data will be collected from diabetic patients 6-15 years old shortly after being diagnosed and compared with results obtained in the healthy group.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Koubek, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. These may be provided upon request.